CLINICAL TRIAL: NCT06362759
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate Quarterly and Monthly TOUR006 in Participants With Chronic Kidney Disease and Elevated High-Sensitivity C-Reactive Protein
Brief Title: A Study to Evaluate TOUR006 in Patients With Chronic Kidney Disease and Elevated Hs-CRP
Acronym: TRANQUILITY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tourmaline Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TOUR006-C01
Record Dates: First submitted 2024-03-27; First posted 2024-04-12 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Chronic Kidney Diseases; Chronic Kidney Insufficiency; Chronic Renal Diseases; Chronic Renal Insufficiency; Kidney Insufficiency, Chronic; C-Reactive Protein; High Sensitivity C-Reactive Protein; Hs-CRP; hsCRP
Keywords: Interleukin-6; IL-6; IL6; Interleukin-6 Inhibitors; Anti-interleukin-6 Agents; Anti-inflammatory Agents; Antiinflammatory Agent; Antiinflammatory Agents; Agents, Antiinflammatory; Anti-inflammatory Agent
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- TOUR006 - 50 MG (Experimental): 50 mg administered subcutaneously at Day 1 and Day 90 (Placebo administered at 30, 60, 120, and 150 Day timepoints)
  Interventions: Drug: TOUR006 - 50 MG
- TOUR006 - 25 MG (Experimental): 25 mg administered subcutaneously at Day 1 and Day 90 (Placebo administered at 30, 60, 120, and 150 Day timepoints)
  Interventions: Drug: TOUR006 - 25 MG
- TOUR006 - 15 MG (Experimental): 15 mg administered subcutaneously at Days 1, 30, 60, 90, 120, and 150
  Interventions: Drug: TOUR006 - 15 MG
- Placebo (Placebo Comparator): Administered subcutaneously at Days 1, 30, 60, 90, 120, and 150
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: TOUR006 - 50 MG — TOUR006 50 MG
  Arms: TOUR006 - 50 MG
Drug: TOUR006 - 25 MG — TOUR006 25 MG
  Arms: TOUR006 - 25 MG
Drug: TOUR006 - 15 MG — TOUR006 15 MG
  Arms: TOUR006 - 15 MG
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study will evaluate the safety, tolerability, pharmacokinetics, and CRP-lowering effect of quarterly and monthly subcutaneous administration of TOUR006 (also known as pacibekitug) in participants with chronic kidney disease and elevated hs-CRP.

DETAILED DESCRIPTION:
Previous clinical studies have suggested that IL-6-driven inflammation plays a key role in the pathogenesis of cardiovascular diseases including atherosclerotic cardiovascular disease (ASCVD) and heart failure. This Phase 2 study will evaluate the safety, tolerability, pharmacokinetics, and CRP-lowering effect of quarterly and monthly subcutaneous administration of TOUR006, a fully human monoclonal antibody against IL-6. TOUR006 binds the IL-6 cytokine and inhibits downstream IL-6 signaling, thereby reducing the pharmacodynamic marker, hs-CRP.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years at time of ICF signature.
* Serum hs-CRP level ≥2.0 mg/L and <15 mg/L
* Diagnosis of chronic kidney disease, eGFR ≥15 and <60 mL/min/1.73 m2 or eGFR ≥60 mL/min/1.73m2 and UPCR>200 mg/g
* Received COVID-19 vaccine at least 30 days prior to the Screening visit, per participant verbal attestation.
* Agreement to comply with contraception and reproduction restrictions

Exclusion Criteria:

* Clinical evidence or suspicion of active infection
* Current or recent COVID-19 infection within 30 days
* Serious infection within 6 months or more than 1 such episode within 18 months
* Any history of a serious opportunistic infection within 18 months
* Known history of immunodeficiency
* History of gastrointestinal ulceration or perforation within 12 months
* History of active diverticulitis, active inflammatory bowel disease, or GI abscess within 12 months
* History of GI bleeding requiring hospitalization and/or transfusion within 6 months
* New York Heart Association Class III or IV congestive heart failure and/or hospitalization for heart failure exacerbation within 6 months
* Acute coronary syndrome, stroke, transient ischemic attack, or other thrombotic or thromboembolic event, or arterial revascularization procedure within 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2025-03-06 (Actual); Study Completion 2025-12-04 (Actual)

PRIMARY OUTCOMES:
Evaluate the effects of TOUR006 compared with placebo on hs-CRP | 90 days
  Evaluates the change from baseline in hs-CRP comparing TOUR006 and placebo

SECONDARY OUTCOMES:
Evaluate the effects of TOUR006 compared with placebo on hs-CRP | 90 days
  Percent of participants achieving hs-CRP less than 2 mg/L
Evaluate the effects of TOUR006 compared with placebo on hs-CRP | 180 days
  Evaluates the change from baseline in hs-CRP comparing TOUR006 and placebo
Evaluate the pharmacokinetics by measuring serum concentrations of TOUR006 | Baseline through Day 365
  Evaluates the serum concentrations of TOUR006 over time
Evaluate the safety and tolerability of TOUR006 in participants with elevated cardiovascular risk and CKD | 365 days
  Evaluates the percentage of participants with treatment emergent adverse events and serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Tourmaline Bio
Locations (38):
- United States (38):
  - Site - 0101, Birmingham, Alabama
  - Site - 0135, Huntsville, Alabama
  - Site - 0145, Huntsville, Alabama
  - Site - 0104, Phoenix, Arizona
  - Site - 0125, San Dimas, California
  - Site - 0112, Valencia, California
  - Site - 0128, Valencia, California
  - Site - 0136, Stamford, Connecticut
  - Site - 0113, Greenacres City, Florida
  - Site - 0149, Pembroke Pines, Florida
  - Site - 0144, Plantation, Florida
  - Site - 0119, Port Orange, Florida
  - Site - 0151, Tampa, Florida
  - Site - 0122, Savannah, Georgia
  - Site - 0106, Chicago, Illinois
  - Site - 0115, Morton, Illinois
  - Site - 0114, Council Bluffs, Iowa
  - Site - 0129, Metairie, Louisiana
  - Site - 0123, Las Vegas, Nevada
  - Site - 0130, Middletown, New York
  - Site - 0110, Charlotte, North Carolina
  - Site - 0117, Fargo, North Dakota
  - Site - 0120, Cincinnati, Ohio
  - Site - 0127, Marion, Ohio
  - Site - 0132, Bethlehem, Pennsylvania
  - Site - 0126, Providence, Rhode Island
  - Site - 0102, Fort Mill, South Carolina
  - Site - 0103, Greenville, South Carolina
  - Site - 0108, Knoxville, Tennessee
  - Site - 0148, Greenville, Texas
  - Site - 0105, Houston, Texas
  - Site - 0111, Lampasas, Texas
  - Site - 0150, McKinney, Texas
  - Site - 0107, San Antonio, Texas
  - Site - 0141, San Antonio, Texas
  - Site - 0109, Manassas, Virginia
  - Site - 0147, Morgantown, West Virginia
  - Site - 0134, Kenosha, Wisconsin